CLINICAL TRIAL: NCT05809102
Title: Results Of Repair Of Flexor Tendon In Zone II Using Minimal Incisions, A Case Series Study
Brief Title: Repair Of Flexor Tendon In Zone II Using Minimal Incisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina S. Fekry, assitant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minimal Incisions in Zone II
Record Dates: First submitted 2023-03-19; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Flexor Tendon Rupture

STUDY DESIGN:
Intervention Model Description: Minimal incisions in repair of Zone II flexor tendon of the hand instead of whole exposure of the tendon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimal incisions (Other): Repair of Zone II using minimal incisions
  Interventions: Procedure: repair of flexor tendon in Zone II

INTERVENTIONS:
Procedure: repair of flexor tendon in Zone II — Repair of Zone II flexor tendon of the hand using minimal incisions instead of whole tendon exposure

SUMMARY:
Repair of the zone II flexor tendon of the hand using minimal incisions is successful with good results which will improve the outcome of the repair.

DETAILED DESCRIPTION:
Flexor tendon laceration in the hand is a common injury with unique characteristics owing to the anatomy of flexor tendons contained within a flexor sheath, requiring good surgical technique as well as strict rehabilitation protocol for regaining function.

The hand is divided into 5 zones (Verdan's). Zone II is described by Bunnel as "No Man's Land" historically back to the 14th century (an area outside London used for executions) because it was previously believed that primary repair should not be done in this zone. After understanding flexor tendon anatomy, biomechanics, and healing new techniques of surgery and anesthesia repair is possible with good results.

Lacerated tendons in zone II can retract proximally to the PIP if the vinculum longus is intact or into the palm if it is disrupted. It will not retract to the level of the wrist because of the origin of the lumbrical insertion into the extensor mechanism.

The laceration can be extended in a Brunner incision or a mid-lateral exposure but it is better skin incisions are minimal to minimize postoperative finger edema, potential adhesions, and injury of any delicate structures.

There are a lot of techniques to retrieve the proximal tendon end as milking, using a hemostat or second incision proximal to the A1 pulley where the tendon is tied to a looped wire of silastic tube and pulled distally through the laceration in the tendon sheath. But little studies discuss the effect of minimal incision on functional outcomes post-operative.

ELIGIBILITY:
Inclusion Criteria:

Age: between 16-60 years.

* Flexor tendon injuries of zone II of any medial four digits in both genders.
* within two weeks.
* Sharp mechanism of injury.
* Single-level injury
* Minimal surgical incision.

Exclusion Criteria:

* Age less than sixteen years old or more than sixty years old.
* Amputation requiring replantation.
* Vascular injury requiring revascularization
* Associated fractures close to the tendon injury.
* Combined flexor and extensor tendon injury.
* Multiple-level injury
* Tendon substance loss
* Insufficient skin and soft tissue coverage.
* Surgical incision for whole tendon exposure.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
range of motions | end point 6 months post-operative
  range of motions of fingers using Jamar finger goniometer

SECONDARY OUTCOMES:
complications | end point 6 months post-operative
  as adhesion formation, which limits active range of motion. joint contracture, tendon rupture, triggering, and pulley failure with tendon bowstringin Infection or neuroma
Healing vs failure of repair | baseline
  questionnaire: can flex finger or not (yes or no)
DASH score using DASH questionnaire | 6 months
  Disabilites of the Arm , Shoulder , Hand score (0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Griffin M, Hindocha S, Jordan D, Saleh M, Khan W. An overview of the management of flexor tendon injuries. Open Orthop J. 2012;6:28-35. doi: 10.2174/1874325001206010028. Epub 2012 Feb 23. PMID 22431948
- [Background] Kotwal PP, Ansari MT. Zone 2 flexor tendon injuries: Venturing into the no man's land. Indian J Orthop. 2012 Nov;46(6):608-15. doi: 10.4103/0019-5413.104183. PMID 23325961
- [Background] Schoffl V, Heid A, Kupper T. Tendon injuries of the hand. World J Orthop. 2012 Jun 18;3(6):62-9. doi: 10.5312/wjo.v3.i6.62. PMID 22720265